CLINICAL TRIAL: NCT05796934
Title: Evaluation of the Moments That Matter Program in Kenya
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Anglican Church of Kenya Development Services - Nyanza (ADS-Nyanza) (Unknown); Episcopal Relief & Development (Unknown)
Responsible Party: Principal Investigator, Joshua Jeong, Research Associate, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB22-1670
Record Dates: First submitted 2023-03-07; First posted 2023-04-04 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Child Development
Keywords: early child development; parenting; Kenya
MeSH Terms: interventions — myotubularin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moments that Matter (Experimental): The intervention group will receive the Moments that Matter (MTM) program, which will involve monthly peer group sessions and monthly home visits that are delivered by ECD promoters over an 18-month program duration, training of faith leaders, and the formation of ECD committees at the community-level.
  Interventions: Behavioral: Moments that Matter (MTM) Program
- Waitlist-Control (No Intervention): The control group will not immediately receive the MTM program but instead the standard of care services (e.g., those provided by community health volunteers which are primarily focused on maternal and child health and nutrition). After follow-up assessments are completed for the trial, then villages in the control group will receive the MTM program.

INTERVENTIONS:
Behavioral: Moments that Matter (MTM) Program — MTM aims to empower caregivers, enhance nurturing care practices, and ultimately improve early child development (ECD). MTM will be targeted to primary caregivers of children aged 0-3 years and implemented over an 18 month period. The primary program delivery agent will be local volunteers ("ECD promoters") who will facilitate monthly peer group sessions and conduct monthly home visits to participants residing in their village. The MTM curriculum covers topics relating to responsive caregiving, early learning, and child security & safety, and gender equality. Faith leaders will also be trained to promote nurturing care and ECD within their sermons and Bible study groups. ECD committees will be also formed among leaders across various sectors (e.g., health, education, faith institutions) to promote nurturing care and ECD at the community level and coordinate MTM activities with program staff, delivery agents, and other existing service providers (e.g., community health volunteers).
  Arms: Moments that Matter

SUMMARY:
This cluster-randomized trial aims to evaluate the impact of the Moments That Matter® (MTM) Program on early child development and caregiving outcomes in two selected counties in western Kenya.

DETAILED DESCRIPTION:
Approximately 43% of children under-5 are at risk of not attaining their developmental potential. Parenting interventions are recommended for improving early childhood development during the earliest years of life. However, there is limited evidence regarding the delivery and effectiveness of parenting interventions to promote early child development outcomes in Kenya specifically. This cluster-randomized trial aims to evaluate the effectiveness of the Moments That Matter® (MTM) Program on early child development and caregiving outcomes in two selected counties in western Kenya. The MTM Program will be implemented by the Anglican Church of Kenya Development Services - Nyanza (ADS-Nyanza), a faith-based organization focused on supporting integrated community-based programs to support the health, wellbeing, and development of the most vulnerable children and families. Various stakeholders - including community volunteers, faith leaders, and ECD committees - will be mobilized and trained to deliver nurturing care and ECD services over an 18-month program period. This trial will enroll primary caregivers of children 0-18 months of age and longitudinally follow the study cohort to ultimately compare changes in early child development and caregiving outcomes between the intervention and waitlist-control study arms. In addition to the impact evaluation, a qualitative implementation evaluation will be conducted to assess quality of delivery, identify factors that influence program effectiveness, and determine program potential for sustainability and scale-up.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver (parent or legal guardian) to a child aged 0-18 months
* Resides in a village selected into the research study
* Caregiver provides informed consent on behalf of both themself and the child to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Early child development | 18 months
  Child development measured using the Caregiver Report of Early Development Index (CREDI) long form version. Scores will be analyzed separately by developmental domain: motor, language, cognitive, and socioemotional development.

SECONDARY OUTCOMES:
Caregiver stimulation practices | 18 months
  Caregiver stimulation practices reported as the number of developmentally-enriching activities that the primary caregiver engaged with the young child (e.g. singing, telling stories). Activities adapted from the Family Care Indicators. A total score will be calculated with higher scores indicated more engagement in stimulation activities.
Home learning materials | 18 months
  Caregiver-reported index of the variety of play and learning materials in the household for child (e.g., home-made toys, store-bought toys, household items). Items adapted from the Family Care Indicators. A total score will be calculated with higher scores indicated more types of home learning materials available for child.
Caregiver disciplinary practices | 18 months
  Caregiver disciplinary practices reported with respect to both harsh punishment (e.g., shook the child, shouted at child) and positive disciplinary practices (e.g., explained why the behavior was wrong) used by the primary caregiver towards the child. Items adapted from Child Discipline Module of Multiple Indicator Cluster Survey. Separate indicators will be created for use of any harsh disciplinary practices or any positive disciplinary practices.
Parenting stress | 18 months
  Parenting distress reported by the primary caregiver using the Parenting Stress Index-Short Form, Parental Distress subscale. Higher total scores indicate greater parenting distress.

OTHER OUTCOMES:
Infant and young child feeding (IYCF) practices | 18 months
  IYCF practices including self-reported breastfeeding and exclusive breastfeeding practices, child dietary diversity score (24 hours), and responsive feeding. Child dietary diversity defined as the number of food groups the child consumed in previous 24 hours based on WHO guidelines. Responsive feeding assessed using a caregiver-reported measure for the style of interaction between primary caregiver and child during mealtime (e.g., talking to child during mealtimes, allowing the child to feed him/herself and explore their food). Higher scores indicate more caregiver responsive feeding behaviors.
Care-seeking for child illness | 18 months
  Indicator for whether primary caregiver sought advice or treatment from appropriate health facility or provider in the event of recent child illness (e.g., cough, fever) based on standard indicator used in UNICEF's Multiple Indicator Cluster Surveys.
Male caregiver involvement | 18 months
  Male caregiver involvement reported by the primary caregivers regarding the number of childcare and household activities performed by the primary male caregiver to support the young child, female partner, or family more broadly (e.g., bathing child, providing money to partner, washing dishes/clothes). Measure developed by authors for this study. Higher scores indicate greater male caregiver involvement.
Gender attitudes | 18 months
  Gender attitudes measured as the primary caregiver's perceptions regarding gender norms and caregiving roles within a household. Items pertain to power dynamics in intimate partner relationships and division of childcare and household responsibilities. Higher scores indicate more gender-equitable attitudes.
Social support | 18 months
  Social support reported by the primary caregiver using the Multidimensional Scale of Perceived Social Support. Higher scores indicate greater perceived social support.
Birth registration | 18 months
  Indicator for whether child's birth was reported by primary caregiver as registered with civil authorities based on standard indicator used in UNICEF's Multiple Indicator Cluster Surveys.
Intimate partner violence | 18 months
  Indicator for whether female primary caregiver reported of any form of intimate partner violence victimization (e.g., physical, emotional) by a male partner using an adapted version of the domestic violence questionnaire from the Demographic and Health Surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Jeong, ScD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Anglican Church of Kenya Development Services - Nyanza, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalam MA, McCann JK, Shakil Z, Gambari A, Ochieng M, Jeong J. Maternal Mental Health and Child Dietary Diversity in Rural Kenya: Findings From a Pooled Analysis of 2 Baseline Studies. Curr Dev Nutr. 2025 Jun 24;9(7):107497. doi: 10.1016/j.cdnut.2025.107497. eCollection 2025 Jul. PMID 40718429